CLINICAL TRIAL: NCT07014462
Title: A Phase 1B Investigator Initiated Study of Safety and Tolerability of Dexamethasone (D) in Combination With Venetoclax-based Low-Intensity Therapy (LIT) in Treatment-Naïve Acute Myeloid Leukemia (AML): DLIT-AML
Acronym: DLIT-AML
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Diego Adrianzen Herrera, Principal Investigator, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003614/UVMC2503
Record Dates: First submitted 2025-05-06; First posted 2025-06-11 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: AML - Acute Myeloid Leukemia
Keywords: AML; Dexamethasone; Venetoclax-
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with ND-AML (Experimental): This is a single-arm, phase 1b, investigator-initiated study evaluating the safety and tolerability of adding dexamethasone to standard venetoclax-based low-intensity therapy (LIT) regimens in treatment-naïve adult patients with acute myeloid leukemia (AML) who are unfit for intensive chemotherapy induction. Participants will receive venetoclax in combination with a hypomethylating agent (azacitidine or decitabine) or low-dose cytarabine, per treating physician's choice. Dexamethasone will be administered orally at 10 mg twice daily on days 1-3 of cycles 1 and 2, and 20 mg once on day 1 of cycles 3 through 6. Treatment will continue for up to 6 cycles (28 days each). The study also includes assessments of patient-reported outcomes and exploratory efficacy endpoints.
  Interventions: Drug: Dexamethasone plus Venetoclax-based Low-Intensity Therapy

INTERVENTIONS:
Drug: Dexamethasone plus Venetoclax-based Low-Intensity Therapy — Participants will receive standard low-intensity therapy (LIT) regimens for newly diagnosed AML, which may include venetoclax combined with either azacitidine, decitabine, or low-dose cytarabine, per treating physician's discretion. In addition, participants will receive dexamethasone administered orally at 10 mg twice daily on days 1-3 of cycles 1 and 2, and 20 mg orally on day 1 of cycles 3 through 6. This intervention is being studied to evaluate whether the addition of dexamethasone improves tolerability and clinical outcomes in patients unfit for intensive chemotherapy.

SUMMARY:
This study is investigating whether adding dexamethasone, an anti-inflammatory medication, to a standard venetoclax-based low-intensity therapy (LIT) is safe and well-tolerated in patients with newly diagnosed Acute Myeloid Leukemia (AML) who are not eligible for intensive chemotherapy.

Study Goals Primary Goal: To assess the safety and tolerability of dexamethasone in combination with venetoclax-based LIT.

Secondary Goal: To evaluate how this treatment affects patients' quality of life using surveys.

Exploratory Goal: To measure the treatment response, including remission rates and signs of minimal residual disease.

What Happens in the Study? Patients will receive treatment over six cycles. Dexamethasone is given in different doses during the first six cycles along with venetoclax and another standard chemotherapy drug.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

ECOG performance status ≤2

Newly diagnosed AML morphologically confirmed in a bone marrow biopsy and aspiration done within 2 months of study enrollment, following the WHO 2022 morphologic classification for myeloid malignancies9

No prior AML treatment (treatment-naïve)

Ineligibility or unwillingness to undergo high-dose chemotherapy induction. Patient candidacy for high dose intensive chemotherapy or ineligibility due to older age or unfit medical status will be determined by the primary treating physician.

Adequate renal function including creatinine clearance > 30 ml/min based on the Cockcroft-Gault equation

Normal liver function with direct bilirubin ≤ 2xULN, ALT and AST ≤ 3xULN, unless deemed to be related to underlying leukemia

Women of child-bearing potential and men (except if previous vasectomy) must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 90 days after completion of therapy

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Ability to understand and the willingness to sign a written informed consent.

Patients with known previous exposure to HMA or LDAC for treatment of a pre-leukemic condition including myelodysplastic syndromes or myeloproliferative neoplasms are eligible.

Exclusion

Acute promyelocytic leukemia diagnosis

Bone marrow transplant expected after first or second cycle of venetoclax-based LIT.

White Blood Cell (WBC) count >25K. If WBC is >25K in an otherwise eligible patient, the use of cytoreduction is allowed and patients can be included when WBC <25K. Hydroxyurea (at any dose) and/or one dose of cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy

The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions: 1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia, or 2) cytoreduction as point 3.2.3.

Uncontrollable infectious disease within 7 days of study enrollment defined as infection confirmed on laboratory tests or imaging and associated with systemic inflammatory response syndrome (SIRS), circulatory compromise or respiratory failure, where steroid treatment may be detrimental according to investigator. Clinically stable febrile neutropenia attributable to AML is not an exclusion criteria.

Patients with any concurrent uncontrolled clinically significant medical condition, laboratory abnormality, or psychiatric illness, which could place the patient at unacceptable risk of study treatment.

Baseline high-dose steroid treatment at dose preceding AML diagnosis for any cause, including concomitant autoimmune disease. The maximum acceptable daily steroid dose is the equivalent of 5 mg of prednisone.

Adrenal insufficiency

Active peptic ulcer disease (PUD), defined as actively having severe pain requiring intervention or bleeding. A simple history of PUD is not an exclusion criterion. If a patient with history of PUD is enrolled, proton pump inhibitor prophylaxis will be used.

Known active hepatitis B (HBV) or Hepatitis C (HCV) infection or known uncontrolled HIV infection. Patients with a history of treated HBV or HCV which has been previously treated, or those with controlled HIV on treatment are eligible.

Patients receiving any other investigational agents

Pregnant or nursing patients

Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications

Patients with uncontrolled diabetes, defined as hemoglobin A1C (HgbA1C) levels >9 and significant baseline hyperglycemia. Patients with controlled diabetes are eligible provided they continue with their treatments and HgbA1C is monitored every 3 months. HgbA1C levels are required only in diabetic patients riteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of adding dexamethasone to venetoclax-based low-intensity therapy in treatment-naïve AML patients | From start of treatment through completion of 6 cycles (each cycle is 28 days; approximately 6 months total)
  The primary outcome will assess the safety and tolerability of the combined regimen. This will include the incidence and severity of adverse events (AEs) graded by NCI CTCAE v5.0, with special attention to clinically significant non-hematologic grade 4 AEs during the first 2 cycles. Overall AE frequency, organ system affected, and hematologic vs. non-hematologic classification will be recorded. Short-term toxicity will be reviewed after enrollment of the first 8-10 patients to determine feasibility for continued accrual.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized patient related data will be incorporated into publications and will be made available to other investigators at reasonable request.